CLINICAL TRIAL: NCT06804343
Title: First Aid Needs of Female Agricultural Workers and the Impact of Basic First Aid Training on Their Knowledge Levels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HaliçÜ-HEM-DR-E-53938333
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: First Aid; Agricultural Workers' Health
Keywords: agricultural worker; woman; first aid; knowledge level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- female agricultural workers (Other): A behavioral intervention consisting of first aid training for female agricultural workers, with a pre-test administered prior to the training, a post-test immediately following the training, and a follow-up test conducted after six months to assess knowledge retention and the application of skills.
  Interventions: Behavioral: first aid training

INTERVENTIONS:
Behavioral: first aid training — A pre-test will be applied to the participants in a single group before the training. After the training is applied, a post-test will be done and a follow-up will be done at the end of 6 months and a post-test will be applied.

SUMMARY:
This study aims to investigate occupational health risks faced by female agricultural workers and their need for first aid training. The objective is to evaluate the effectiveness of a basic first aid training program in enhancing knowledge and practical skills, thereby improving workplace safety and individual health outcomes.

DETAILED DESCRIPTION:
This research focuses on identifying the first aid needs of female agricultural workers and assessing the impact of a structured basic first aid training program on their knowledge and practical skills. The study will be conducted in Kadıköy neighborhood, Silivri district, Istanbul Province, a region with active agricultural activities.

The training program integrates theoretical and practical components, designed in collaboration with 10 experts in the field. Theoretical sessions will be delivered through presentations and educational brochures. Practical training will include hands-on demonstrations and skill assessments, focusing on bleeding control and the Heimlich maneuver. Simulated scenarios will be employed using an arm model with moulage and a CPR manikin, with performance evaluated through standardized assessment forms.

The study is scheduled to take place from November 2024 to May 2025. Data collection will involve pre-training assessments to establish baseline knowledge and skills, immediate post-training evaluations to determine the program's effectiveness, and a six-month follow-up to assess knowledge retention and the real-world application of first aid skills. A total of 43 participants, calculated using G*Power analysis for a repeated-measures design, will ensure adequate statistical power.

By addressing the first aid needs of female agricultural workers, this study aims to enhance workplace safety, empower workers to manage occupational risks effectively, and contribute to better health outcomes within agricultural settings.

ELIGIBILITY:
Inclusion Criteria:

* Being a female agricultural worker,
* Being 18 years of age or older,
* Willing to participate in the study,
* Having no hearing impairment.

Exclusion Criteria:

• Not having attended one of the training sessions conducted by the instructor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female agricultural worker
Enrollment: 43 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
The Impact of Basic First Aid Training on Knowledge Levels | The initial assessment will be conducted immediately after training, followed by a six-month evaluation.
  The primary outcome of this study is to assess the effect of basic first aid training on the knowledge levels and practical skills of female agricultural workers, both prior to and following the training. The evaluation will focus on meaningful improvements in knowledge and practical skills, which will be measured using the 'First Aid Knowledge Level Survey' and 'Practical Skills Assessments.' The practical skills assessments will involve evaluating the ability to apply bandages in cases of bleeding and to perform the Heimlich maneuver for airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel ERKAL İLHAN, Prof.Dr., Study Director — Haliç University
Locations (1):
- İstanbul Silivri İlçesi Kadıköy Mahallesi Muhtarlığı, Istanbul, Silivri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Once the study data are collected, including distribution demographics, baseline measurements, and outcomes, they will be shared following publication of the trial results.
Supporting Information: SAP, CSR
Time Frame: It starts with the publication, there is no end date
Access Criteria: Only sharing data will be possible if an independent review confirms the methods used to ensure that the analyses are valid and reliable. The data to be shared must fully comply with ethical, legal and scientific requirements. In addition, requests for data sharing must include a proposal for the purpose of use and analysis, in accordance with mathematical powers. Data will only be shared for use in a manner that protects confidentiality and complies with ethical rules.